CLINICAL TRIAL: NCT06198907
Title: A Phase 2, Open-label, Single Arm Study to Investigate the Safety and Efficiency of Golidocitinib in Combination With Sintilimab in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) With PD-L1TPS ≥ 1%)
Brief Title: Golidocitinib in Combination With Sintilimab for PD-L1 Selected Treatment Locally Advanced or Metastatic Non-Small Cell Lung Cancer(NSCLC)
Acronym: JACKPOT33
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Dizal Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Jie Wang, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZ2023J0002
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A Dose escalation (Experimental): Dose escalation part Golidocitinib in combination with sintilimab
  Interventions: Drug: Golidocitinib; Drug: Sintilimab
- Part B Dose expansion cohort 1 (PD-L1 TPS ≥ 50%) (Experimental): Dose expansion cohort 1, Golidositinib plus Sintilimab following Sintilimab
  Interventions: Drug: Golidocitinib; Drug: Sintilimab
- Part B Dose expansion cohort 2 (PD-L1 TPS 1-49%) (Experimental): Dose expansion cohort 2, Golidositinib plus Sintilimab following Sintilimab + chemotherapy
  Interventions: Drug: Golidocitinib; Drug: Sintilimab; Drug: platinum doublet chemotherapy

INTERVENTIONS:
Drug: Golidocitinib — Daily dosing of golidocitinib
Drug: Sintilimab — Sintilimab, 200mg, intravenous, every 3 weeks.
Drug: platinum doublet chemotherapy — Pemetrexed or nab-paclitaxel +carboplatin, intravenous, every 3 weeks for 2 cycles
  Arms: Part B Dose expansion cohort 2 (PD-L1 TPS 1-49%)

SUMMARY:
This is a phase 2 Study to investigate the safety, tolerability, and anti-tumor activity of golidocitinib in combination with sintilimab as the front-line treatment for patients with metastatic PD-L1 positive non-small cell lung cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide a signed and dated, written informed consent.
2. Adults aged ≥18 to 75 years.
3. ECOG performance status 0-1.
4. Predicted life expectancy ≥ 12 weeks
5. Histologically or cytologically confirmed non-small-cell lung cancer (NSCLC) , Stage IIIB/IIIC (not suitable for concomitant chemoradiotherapy) or Stage IV according to AJCC 8th
6. Without EGFR or ALK mutations.
7. Adequate bone marrow reserve and organ system functions.
8. Patients with stable and symptomatic brain metastasis (BM) can be enrolled.

Part A Dose escalation:

Patients must have relapsed after or been refractory/intolerant to ≥ 1 prior systemic therapy(ies) for NSCLC

Part B dose expansion:

1. At least one measurable lesion according to RECIST 1.1.
2. Previously systemic untreated for advanced disease.
3. PD-L1 TPS ≥ 50% (cohort 1), PD-L1 TPS 1-49% (cohort 2)

Exclusion Criteria:

1. Histopathology confirmed a mixture of NSCLC and small-cell lung cancer
2. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
3. Prior malignancy within 5 years
4. History of organ transplantation or hematopoietic stem cell transplantation
5. Sever lung function decline or interstitial lung disease that has required oral or IV steroids
6. Active autoimmune disease requiring systemic therapy within 2 years
7. Immunodeficiency, or being treated with immunosuppressive therapy (including systemic glucocorticoid) within 7 days prior to the first dose of study treatment.
8. Active infections
9. Significant cardiac disorder
10. Other serious or uncontrolled systemic diseases assessed by the investigator.

Part A Dose escalation:

1. Prior systemic therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or stimulatory or synergistic T-cell receptor (CTLA-4、OX-40、CD137) within 4 weeks

Part B Dose Expansion:

1. Any prior systemic anti-tumor therapy
2. Prior systemic immunotherapy, including anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or stimulatory or synergistic T-cell receptor (CTLA-4、OX-40、CD137)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 69 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) (cohort1) | through study completion, an average of 1 year
  Complete response (CR) or partial response (PR) per investigator assessment according to RECIST 1.1
Progression-free survival (PFS) (cohort2) | through study completion, an average of 1 year
  Time from first administration of study drug to first documented disease progression or death per investigator assessment according to RECIST 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | through study completion, up to 36 months
  time from first administration of study drug to death
Incidence of Adverse Events | through study completion, up to 36 months
  Frequency an severity of AEs according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, MD,PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No